CLINICAL TRIAL: NCT00952042
Title: Heavy Slow Resistance Versus Eccentric Training in the Treatment of Achilles Tendinopathy. A Randomized Controlled Trial.
Brief Title: Resistance Training as Treatment of Achilles Tendinopathy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Copenhagen (Other)
Responsible Party: Principal Investigator, Rikke Beyer, Phd. stud. Rikke Beyer, University of Copenhagen
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Kongsgaard2
Record Dates: First submitted 2009-08-03; First posted 2009-08-04 (Estimated); Last update posted 2014-07-21 (Estimated); Status verified 2014-07

CONDITIONS: Achilles Tendinopathy
Keywords: Tendinopathy, Achilles, Eccentric training, Heavy slow resistance training
MeSH Terms: conditions — Tendinopathy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Heavy slow resistance training (Experimental): 12 wks of heavy slow resistance training. training three times per week. each session: 3 heel-raise exercises. 12-6RM. Slow contractions.
  Interventions: Other: Heavy slow resistance training
- Eccentric resistance training (Active Comparator): 12 wks of eccentric resistance training. 3 x 15 Eccentric heel-raises performed twice daily.
  Interventions: Other: Eccentric resistance training

INTERVENTIONS:
Other: Heavy slow resistance training — Heel-raises. 12-6RM. each contraction performed slowly. three times weekly for 12 weeks
  Arms: Heavy slow resistance training
Other: Eccentric resistance training — Eccentric heel-raises. 3 x 15 reps performed twice daily for 12 wks.
  Arms: Eccentric resistance training

SUMMARY:
The use of eccentric resistance training as management of Achilles tendinopathy is widespread. The investigators have recently demonstrated that heavy slow resistance training was superior in the management of patellar tendinopathy.

Hypothesis: heavy slow resistance training is more effective than eccentric resistance training in the clinical management of Achilles tendinopathy.

ELIGIBILITY:
Inclusion Criteria:

* Unilateral Achilles tendon pain,
* Symptoms for at least three months,
* Ultrasonographical tendon abnormalities, AND
* Able to comply with both intervention arms.

Exclusion Criteria:

* Bilateral symptoms,
* Previous surgery below knee,
* Corticosteroid injections below the knee during past year,
* Hypercholesterol,
* Diabetes, OR
* Arthritis.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 47 (Actual)
Dates: Start 2009-07; Primary Completion 2012-10 (Actual); Study Completion 2012-10 (Actual)

PRIMARY OUTCOMES:
VISA-A score | 0,12 wks + 1yr follow-up

SECONDARY OUTCOMES:
Tendon thickness | 0,12 wks + 1yr follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Rikke Beyer, PhD. stud, Principal Investigator — Institute of Sports Medicine Copenhagen (www.ismc.dk)
Locations (1):
- Institute of Sports Medicine Copenhagen. Bispebjerg Hospital, Copenhagen NV, Denmark

REFERENCES:
- See also: Related Info — http://ismc.dk